CLINICAL TRIAL: NCT01029288
Title: Impact of Decision Aids to Enhance Shared Decision Making for Diabetes
Acronym: DAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DK084009
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
Keywords: Diabetes; Decision aid; Cardiovascular risk; Patient education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin Choice Decision Aid (Active Comparator): Subjects will receive an intervention of Statin Choice Decision Aid and usual care for antihyperglycemic medication discussion with their clinician.
  Interventions: Other: Statin Choice Decision Aid; Other: Usual care for antihyperglycemic medication
- Diabetes Medication Choice Decision Aid (Active Comparator): Subjects will receive an intervention of Diabetes Medication Choice Decision Aid and usual care for lipid therapy medication discussion with their clinician.
  Interventions: Other: Diabetes Medication Choice Decision Aid; Other: Usual care for lipid therapy medication

INTERVENTIONS:
Other: Diabetes Medication Choice Decision Aid — Diabetes Medication Choice cards
  Arms: Diabetes Medication Choice Decision Aid
Other: Statin Choice Decision Aid — Statin Choice Cards
  Arms: Statin Choice Decision Aid
Other: Usual care for lipid therapy medication — Clinicians will follow their clinic's usual care practice for lipid therapy medication (statin) discussions.
  Arms: Diabetes Medication Choice Decision Aid
Other: Usual care for antihyperglycemic medication — Clinicians will follow their clinic's usual care practice for antihyperglycemic medication discussions.
  Arms: Statin Choice Decision Aid

SUMMARY:
The proposed trial seeks to determine the impact of patient decision aids versus usual care on measures of patient involvement in decision-making, diabetes care processes, medication adherence, glycemic and cardiovascular risk factor control, and resource utilization in nonurban practices in the Midwestern United States. Upon completion of this trial, the investigators will have new knowledge about both the effectiveness of diabetes decision aids in nonacademic nonurban practices and about the processes that promote or inhibit the successful implementation of patient decision aids in such practices.

DETAILED DESCRIPTION:
Type 2 diabetes causes loss of quality and diminished duration of life for over 24 million Americans with great costs and heavy burden of treatment for both society and for affected families. Decision aids are tools that help clinicians involve patients in making deliberate choices by providing accessible information about the options available and their outcomes. We propose to conduct a cluster randomized trial to obtain an estimate of the impact of patient decision aids versus usual care on measures of patient involvement in decision making, diabetes care processes, medication adherence, glycemic and cardiovascular risk factor control, and resource utilization.

Participating clinicians will be trained to use decision aid tools to discuss starting either new diabetes medications or new statins with their enrolled patients. Surveys completed by clinicians and patients will assess satisfaction with decision making and knowledge gained by patients. 3- and 6-month follow-up surveys completed by patients will assess adherence to chosen medications and sustained knowledge. Primary analysis will be conducted utilizing generalized linear models. Some visits will be video and/or audio recorded with permission, and a small subset of patients, clinicians, and support staff will be interviewed by an experienced qualitative researcher using a semi-structured interview guide.

Primary care practices were enrolled then matched by size (less than or equal to 2 clinicians or greater than 2 clinicians) and randomly allocated by a statistician to 1) the use of the Diabetes Medication Choice decision aid and usual care for lipid therapy medication (statin) discussion during the encounter with subjects or to 2) the use of the Statin Choice decision aid and usual care for antihyperglycemic mediations discussion during the encounter with subjects.

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider is participating in trial
* Are an adult (≥ 18 years) with type 2 diabetes
* English speaking
* Recognize their primary care provider as their main diabetes care provider
* Declare being available for follow-up for six months after treatment decision

Exclusion Criteria:

- Have major barriers to provide written informed consent and to participate in shared decision making (i.e., severe vision or hearing impairment, cognitive impairment, non-English speaking)

Additional Inclusion Criteria for Diabetes Medication:

* Have a clinical diagnosis of type 2 diabetes for one year or more (c-peptide test is not required)
* Use 0, 1, or 2 oral hypoglycemic agents at maximum doses
* Have stable but inadequate glycemic control or worsening glycemic control as identified by their most recent HbA1c measure (within 12 months of the time of eligibility over 7.3%
* Be identified by provider as a medically-appropriate candidate for diabetes medications, (i.e., have not contraindications to taking the medications, e.g., allergy).

Additional Exclusion Criteria for Diabetes Medication:

- Use insulin therapy.

Additional Inclusion Criteria for Cardiovascular Medication:

* Have a clinical diagnosis of type 2 diabetes for any duration (c-peptide test is not required).
* Be identified by provider as a medically-appropriate candidate for statins, (i.e., have not contraindications to taking the medications, e.g., allergy).

Additional Exclusion Criteria for Cardiovascular Medication:

- Use a statin currently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Decisional quality (knowledge, decisional conflict, and satisfaction) | Immediately (within 10 minutes) following clinical encounter, and 3- & 6-months post encounter

SECONDARY OUTCOMES:
Provider satisfaction | Immediately following clinical encounter
Patient medication adherence | 6-months following clinical encounter

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, M.D., M.Sc., Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - MCHS-Albert Lea, Albert Lea, Minnesota
  - MCHS-Austin, Austin, Minnesota
  - Mayo Family Clinic, Kasson, Minnesota
  - Olmsted Medical Center, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Branda ME, LeBlanc A, Shah ND, Tiedje K, Ruud K, Van Houten H, Pencille L, Kurland M, Yawn B, Montori VM. Shared decision making for patients with type 2 diabetes: a randomized trial in primary care. BMC Health Serv Res. 2013 Aug 8;13:301. doi: 10.1186/1472-6963-13-301. PMID 23927490
- [Derived] Wyatt KD, Branda ME, Inselman JW, Ting HH, Hess EP, Montori VM, LeBlanc A. Genders of patients and clinicians and their effect on shared decision making: a participant-level meta-analysis. BMC Med Inform Decis Mak. 2014 Sep 2;14:81. doi: 10.1186/1472-6947-14-81. PMID 25179289
- [Derived] Ruud KL, Leblanc A, Mullan RJ, Pencille LJ, Tiedje K, Branda ME, Van Houten HK, Heim SR, Kurland M, Shah ND, Yawn BP, Montori VM. Lessons learned from the conduct of a multisite cluster randomized practical trial of decision aids in rural and suburban primary care practices. Trials. 2013 Aug 21;14:267. doi: 10.1186/1745-6215-14-267. PMID 23965227
- [Derived] Tiedje K, Shippee ND, Johnson AM, Flynn PM, Finnie DM, Liesinger JT, May CR, Olson ME, Ridgeway JL, Shah ND, Yawn BP, Montori VM. 'They leave at least believing they had a part in the discussion': understanding decision aid use and patient-clinician decision-making through qualitative research. Patient Educ Couns. 2013 Oct;93(1):86-94. doi: 10.1016/j.pec.2013.03.013. Epub 2013 Apr 15. PMID 23598292
- See also: Related Info — http://kercards.e-bm.info